CLINICAL TRIAL: NCT04782349
Title: Additive Effect of Mulligan Mobilization With Low Level Laser Therapy for Treatment of Patients With Shoulder Adhesive Capsulitis: Double Blinded, Randomized Controlled Trial.
Brief Title: Mulligan Mobilization With Laser for Shoulder Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment of frozen shoulder
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2021-03

CONDITIONS: Shoulder Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Low-Level Light Therapy; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high intensity laser group (Experimental)
  Interventions: Other: mulligan mobilization with low level laser therapy and traditional physical therapy exercises
- low intensity laser group (Experimental)
  Interventions: Other: low level laser therapy and traditional physical therapy exercises
- control group (Other)
  Interventions: Other: physical therapy exercises

INTERVENTIONS:
Other: mulligan mobilization with low level laser therapy and traditional physical therapy exercises — for mulligan mobilization: for improving the limited range of motion of shoulder joint, the therapist will apply posterolateral mobilization for the shoulder joint. Three sets of painless glides of 10 repetitions will be applied with a rest interval of 30 s between each set.
  For low level laser application: Laser specifications is as follows: 850 nm wave length and pulsed application with 8 W applied for 20 minutes. laser will be applied over painful points of the shoulder.
  For traditional physical therapy exercises: the patients will receive the following exercise program: self stretching exercises for shoulder joint, pully exercises, back climbing exercises, finger ladder exercises, circumduction exercises and pendulum exercises
  Arms: high intensity laser group
Other: low level laser therapy and traditional physical therapy exercises — patients in this group will receive low level laser and traditional physical exercises as described before for group (A)
  Arms: low intensity laser group
Other: physical therapy exercises — The patients will receive traditional physical therapy exercises only as described before for group (A)
  Arms: control group

SUMMARY:
Adhesive capsulitis (frozen shoulder) is a condition of uncertain etiology characterized by pain and progressive loss of both active and passive shoulder motion.

Shoulder pain and stiffness are accompanied by disability. It is thought that the incidence is 3 to 5% in the general population. Laser therapy is widely used for treating different musculoskeletal diseases, because of its ability to reduce pain and improve the physical function. Also, MWM when used for shoulders with limited range of motion because of pain had shown improvement in range of motion and pressure pain threshold. Previous studies have investigated the efficacy of combining different manual technique with LLLT for treating pain in some body parts. However, up till now the combined effect of MWM with LLLT for treatment of patients with shoulder adhesive capsulitis have not been investigated.

So, the present randomized controlled study will be conducted to investigate the effect of adding mulligan mobilization with movement to low level laser therapy in treatment of patients with shoulder adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* The participant selected for the study were patients (both male and female).
* Subjects diagnosed diagnosed by physicians with Magnetic Resonance Imaging (MRI).

  & referred by an Orthopedician with stage 2 Adhesive Capsulitis.
* Age group of 40-60 years of old.
* painful condition of at least 3 months with 50% restriction in passive shoulder flexion, abduction and external rotation, in a sagittal plane compared with opposite side.
* The severity of pain on visual analogue scale was higher than three out of ten, pain aggravated by movements.
* patients were suffering from pain and limitation in the motion for more than 3 month.

Exclusion Criteria:

* Patients with any shoulder injury or trauma, surgical release of capsule.
* Previous manipulation done under anaesthesia of the affected shoulder in the preceding 4 weeks.
* Other conditions involving the shoulder (eg. rheumatoid arthritis, osteoarthritis, damage of the glenohumeral cartilage, osteoporosis, or malignancies in the shoulder region).
* Pain or disorders of the cervical spine, elbow, wrist, or hand.
* Presence of medical conditions such as cardiac disease, infections, coagulation disorder.
* patients having any intra articular injection, or physiotherapy treatment in the affected shoulder during the last three months.
* patients with musculoskeletal disorder (any type of fracture), any history of surgery on that shoulder and patients with tendon calcification, patients with cervical rib, rotator cuff tear patients.
* Patients have insulin-dependent diabetes mellitus.
* Bilateral Frozen Shoulder
* systemic inflammatory joint disease (such as rheumatoid arthritis or polymyalgia rheumatica).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | change from base line at three weeks
  Pain intensity will be measured with Visual Analog Scale (VAS). The patient will be asked to mark the severity of pain on a 100-mm line with "no pain" on one end and "most unbearable pain" on the other end

SECONDARY OUTCOMES:
pain pressure threshold | change from baseline at three weeks
  - The most sensitive point will be located over the anterior aspect of the shoulder by manual palpation and will be marked with a permanent marker so that the same point could be used for pre- and post-condition application measures. This process will be repeated three times with a 30-s rest period between each measurement.
Shoulder range of motion (flexion, abduction, and external rotation) | change from baseline at three weeks
  A universal goniometer will be used to measure the ROM.
  * patient in supine lying with shoulder neutral.
  * Flexion ROM will be measured with the stationary arm of goniometer parallel to the trunk, and the moving arm parallel with the affected arm. Fulcrum will be placed in the point of lateral aspect of acromion process.
  * For measurement of shoulder abduction, the fulcrum of the goniometer will be placed anterior to acromion process, stationary arm parallel to midline of sternum and movable arm will be placed at the midline of humerus. The patient is asked to abduct the arm as much as possible and the reading of the goniometer will be noted.
  * For external rotation of the shoulder, patient is positioned in supine lying and arm abducted to 90 degree and elbow at 90 degree. Fulcrum of goniometry over olecranon and stationary arm perpendicular to floor, moving arm is aligned parallel to the ulna. The patient is asked to rotate externally as much as possible.
Disability of Arm Shoulder Hand (DASH): | change from baseline at three weeks
  - The functional index designed to determine the symptoms and limitations that participant was experiencing while performing daily activities. This scale consists of 30 items in the form of activities of daily living with each item scoring from 0 to 4, where 0 is no difficulty in performing that activity and 4 is unable to do that activity. The DASH score is expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

REFERENCES:
- [Background] Lirio Romero C, Torres Lacomba M, Castilla Montoro Y, Prieto Merino D, Pacheco da Costa S, Velasco Marchante MJ, Bodes Pardo G. Mobilization With Movement for Shoulder Dysfunction in Older Adults: A Pilot Trial. J Chiropr Med. 2015 Dec;14(4):249-58. doi: 10.1016/j.jcm.2015.03.001. Epub 2015 Nov 24. PMID 26793036
- [Background] Noten S, Meeus M, Stassijns G, Van Glabbeek F, Verborgt O, Struyf F. Efficacy of Different Types of Mobilization Techniques in Patients With Primary Adhesive Capsulitis of the Shoulder: A Systematic Review. Arch Phys Med Rehabil. 2016 May;97(5):815-25. doi: 10.1016/j.apmr.2015.07.025. Epub 2015 Aug 15. PMID 26284892
- [Background] Ip D, Fu NY. Two-year follow-up of low-level laser therapy for elderly with painful adhesive capsulitis of the shoulder. J Pain Res. 2015 May 25;8:247-52. doi: 10.2147/JPR.S84376. eCollection 2015. PMID 26045677